CLINICAL TRIAL: NCT00814437
Title: Physiological Role of KiSS-1/GPR54 System in the Human Ovary
Acronym: 001-KIS
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Vida Recoletas Sevilla (Other)
Responsible Party: Principal Investigator, Manuel Fernandez-Sanchez, Primary Investigator, Vida Recoletas Sevilla
Other Study IDs: IVISEV-001-KIS
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Human granulosa cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Donors: Oocyte donor

SUMMARY:
The aim of this project is to study the physiological role of the KiSS-1/GPR54 system in the granulosa cells of the human ovary.

ELIGIBILITY:
Inclusion Criteria:

* Consenting oocyte donors

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy oocyte donors
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Fernández-Sánchez, PhD, MD, Principal Investigator — Vida Recoletas Sevilla